CLINICAL TRIAL: NCT00374530
Title: Headache Inducing Characteristics and Possible Changes in Cerebral Blood Flow After Administration of PGE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: KA-20060026
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Dinoprostone

INTERVENTIONS:
Drug: PGE2

SUMMARY:
Before, during and after intravenous administration of PGE2 we score/measure headache, rCBF, blood flow in the middle cerebral artery and diameter of superficial temporal artery and correlate that to known pathophysiology of headache to see if PGE2 is involved in headache pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Primary Headache, headache on the day of the investigation, hypertension, hypotension, pregnant/nursing, daily intake of medication (except oral contraceptives), Cardiovascular or CNS disease, drug/alcohol abuse, psychiatric disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-08

PRIMARY OUTCOMES:
Headache

SECONDARY OUTCOMES:
rCBF, blood flow, diameter of STA/RA, HR, BP

CONTACTS AND LOCATIONS:
Overall Officials: Troels Wienecke, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Glostrup, Denmark